CLINICAL TRIAL: NCT04574375
Title: A Prospective, Observational (Non-interventional), International Study to Assess Effectiveness of Conservative Treatments in Chronic Venous Disease
Brief Title: Chronic VEnous dIsorders maNagement and Treatment effectivenesS evaluaTion in Chronic vEnous Disease, an International Program
Acronym: VEIN STEP
Status: Completed | Type: Observational
Sponsor: Servier Affaires Médicales (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Other Study IDs: DIM-05682-007-INT
Record Dates: First submitted 2020-09-15; First posted 2020-10-05 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2022-12

CONDITIONS: Chronic Venous Disease
Keywords: observationnal; QoL

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of this study is to assess in real-life settings the effectiveness of conservative treatments on symptoms, signs and quality of life, in patients consulting for CVD

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Patient consulting spontaneously or referred for symptomatic venous disorders
* Diagnosis of chronic venous disease according to investigator's judgment

Exclusion Criteria:

* Presence of known severe systemic disease likely to interfere with the study evaluation
* Patients with lower limb arterial disease
* Patient with any other concomitant disease or treatment that may interfere with lower limb pain or edema
* Patient consulting for an emergency not related to venous disease
* Patient currently taking any treatment for chronic venous disorders, either with venoactive drug or with compression hosiery
* Procedure or surgery for venous disease planned during the study
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients consulting spontaneously or referred for symptomatic CVD not requiring surgical treatment
Sampling Method: Non-Probability Sample
Enrollment: 6419 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Global leg symptoms severity | week 4
  Measured by visual analogue scale (VAS) and questioning with 4 points rate
Global improvement | Week 4
  Measured by Patient Global Impression of Change (PGIC) scale, and time to improvement.
Disease severity | Week 4
  Measured by VCSS (Venous Clinical Severity score)
Quality of Life | Week 4
  Measured by CIVIQ-14 questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Servier Affaires Medicales, Suresnes, France

REFERENCES:
- [Derived] Mezalek ZT, Feodor T, Chernukha L, Chen Z, Rueda A, Sanchez IE, Ochoa AJG, Chirol J, Blanc-Guillemaud V, Lohier-Durel C, Ulloa JH. VEIN STEP: A Prospective, Observational, International Study to Assess Effectiveness of Conservative Treatments in Chronic Venous Disease. Adv Ther. 2023 Nov;40(11):5016-5036. doi: 10.1007/s12325-023-02643-6. Epub 2023 Sep 20. PMID 37728696
- See also: Publication with results from MORROCO — https://www.phlebolymphology.org/vein-step-chronic-venous-disorders-management-and-treatment-effectiveness-evaluation-in-chronic-venous-disease-an-international-observational-prospective-study-results-from-morocco/
- See also: VEIN STEP: A Prospective, Observational, International Study to Assess Effectiveness of Conservative Treatments in Chronic Venous Disease (in Advances in Therapy, September 2023) — http://link.springer.com/article/10.1007/s12325-023-02643-6